CLINICAL TRIAL: NCT00782171
Title: Immediate and Delayed Loading of 4.1 mm and 4.8 mm Implants in the Posterior Mandible & Maxilla: A Controlled Randomized Study of Single or 2-4 Unit Restorations Loaded Immediately After Surgery or Four Weeks After Surgery
Brief Title: Evaluation of Immediate Versus Delayed Loading of Dental Implants With a Modified Surface
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Institut Straumann AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR 06/03
Record Dates: First submitted 2008-10-28; First posted 2008-10-31 (Estimated); Results first posted 2017-06-20 (Actual); Last update posted 2017-06-20 (Actual); Status verified 2017-04

CONDITIONS: Partial Edentulism
Keywords: Dental implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immediate Loading (Active Comparator): SLActive dental implant(s) will be restored with a temporary restoration on the day of surgery.
  Interventions: Device: SLActive dental implant
- Early Loading (Active Comparator): Healing caps will be placed on the SLActive dental implant(s) immediately after surgery. A provisional restoration will be placed between day 28 to day 34 post surgery
  Interventions: Device: SLActive dental implant

INTERVENTIONS:
Device: SLActive dental implant — Straumann® SLActive implants will be placed. Implants in Arm 1 will be restored with a temporary restoration on the day of surgery.
  Implants in Arm 2 will receive healing caps immediately after surgery and a provisional restoration will be placed between day 28 to day 34 post-surgery.
  In both arms, the final restoration will be placed between 140 and 160 days (20 to 23 weeks) post-surgery.
  Other Names: SLActive

SUMMARY:
The purpose of this study is to evaluate the performance of a new dental implant with a modified surface in different loading protocols.

DETAILED DESCRIPTION:
This study is a post-market randomized study whereby each patient will receive 1 to 4 implants placed in the posterior maxilla or mandible. The primary objective of this randomized open study is to evaluate the performance in immediate and delayed loading (4 weeks) of Straumann standard solid screw 4.1mm and the 4.8 mm diameter wide neck implants with a new surface. These implants will support single crowns or 2 to 4 unit bridge restorations in the posterior maxilla or mandible and the treatment will be evaluated for the immediate and delayed loading procedures at one year post surgery. Patients will be allocated into two groups and then randomized into immediate or delayed loading arms.

ELIGIBILITY:
Inclusion Criteria:

* Males and females must be at least 18 years of age
* Have at least one missing tooth in positions FDI 4, 5, 6, or 7 in any quadrant (ADA positions 2, 3, 4, 5; or 12, 13, 14, 15; or 20, 21, 22, 23; or 28, 29, 30, 31.)
* Subjects desire an implant supported restoration on1 to 4 implants per quadrant
* The tooth/teeth position(s) at the proposed implant site must have been extracted or lost at least 4 months before the date of implantation and be fully healed
* Adequate bone quality and quantity at the implant site to permit the insertion of a Straumann standard 4.1 mm diameter implant of at least 8 mm length without the use of concurrent bone augmentation techniques. If more bone is available and is indicated a Straumann standard 4.8 mm diameter implant with a wide neck of at least 8 mm length may be used, i.e. implant insertion sites must have sufficient bone height such that the implant will not encroach on vital structures and sufficient width that a minimum of 1 mm of bone lingual and buccal bone will remain
* The opposing dentition must be natural teeth or fixed crowns or bridges on natural teeth or implants. Removable prostheses or dentures opposing the study implants are not allowed
* Patients must be committed to the study for its full duration.

Exclusion Criteria:

* Presence of conditions requiring chronic routine prophylactic use of antibiotics (e.g., history of rheumatic heart disease, bacterial endocarditis, cardiac valvular anomalies, prosthetic joint replacements)
* Medical conditions requiring prolonged use of steroids
* History of leukocyte dysfunction and deficiencies
* History of bleeding disorders
* History of neoplastic disease requiring the use of chemotherapy
* History of radiation therapy to the head and neck
* Patients with history of renal failure
* Patients with severe or uncontrolled metabolic bone disorders
* Uncontrolled endocrine disorders
* Physical handicaps that would interfere with the ability to perform adequate oral hygiene
* Use of any investigational drug or device within the 30 day period immediately prior to implant surgery on study day 0
* Alcoholism or drug abuse
* Patients infected with HIV
* Patients who smoke >10 cigarettes per day or cigar equivalents, or who chew tobacco
* Conditions or circumstances, in the opinion of the investigator, which would prevent completion of study participation or interfere with analysis of study results, such as history of non-compliance, or unreliability
* Local inflammation, including untreated periodontitis
* Mucosal diseases such as erosive lichen planus
* History of local irradiation therapy
* Presence of osseous lesions
* Unhealed extraction sites (less than 4 months post extraction of teeth in intended sites)
* Bone surgery (bone grafts, guided tissue regeneration techniques for bone enhancement) prior to implant placement unless performed more than 6 months prior to implant placement and the site fully healed. Note: Minor bone enhancement using harvested bone from the implant site and a resorbable membrane is allowed at the time of implant placement
* Patients requiring bone grafting at the surgical sites at the time of surgery.
* Severe bruxing or clenching habits
* Persistent intraoral infection
* Lack of primary stability of one (or more) implant(s) at surgery. In this instance the patient must be withdrawn and the patient treated accordingly
* Patients with inadequate oral hygiene or unmotivated for adequate home care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Actual)
Dates: Start 2004-07; Primary Completion 2006-10 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Axel Zöllner, DDS, Principal Investigator — Private Universität Witten/ Herdecke
Locations (19):
- United States (3):
  - Private Practice, Boca Raton, Florida
  - Private Practice, Indianapolis, Indiana
  - University of Pennsylvania, Philadelphia, Pennsylvania
- Tiroler Landeskrankenanstaltengesellschaft mbH, Innsbruck, Austria
- Germany (5):
  - Praxisklinik fur Mund- Keifer- und Gesichtschirurgie, Bochum
  - Private Practice, Fürth
  - Klinikum Nord-Heidberg, Hamburg
  - Private Practice, Weiden
  - Private Universitat Witten, Witten
- Ireland (2):
  - Queens University, Belfast
  - Dublin Dental Hospital, Dublin
- Rijnland Hospital, Leiderdorp, Netherlands
- Portugal (2):
  - Faculdade de medicina de coimbra, Coimbra
  - Private Practice, Porto
- Spain (3):
  - Private Practice, Barcelona
  - Private Practice, Málaga
  - Clinica Periobalear, Palma de Mallorca
- Private Practice, Falun, Sweden
- Private Practice, Sankt Gallen, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zollner A, Ganeles J, Korostoff J, Guerra F, Krafft T, Bragger U. Immediate and early non-occlusal loading of Straumann implants with a chemically modified surface (SLActive) in the posterior mandible and maxilla: interim results from a prospective multicenter randomized-controlled study. Clin Oral Implants Res. 2008 May;19(5):442-50. doi: 10.1111/j.1600-0501.2007.01517.x. PMID 18416725
- [Result] Ganeles J, Zollner A, Jackowski J, ten Bruggenkate C, Beagle J, Guerra F. Immediate and early loading of Straumann implants with a chemically modified surface (SLActive) in the posterior mandible and maxilla: 1-year results from a prospective multicenter study. Clin Oral Implants Res. 2008 Nov;19(11):1119-28. doi: 10.1111/j.1600-0501.2008.01626.x. PMID 18983314
- [Result] Nicolau P, Korostoff J, Ganeles J, Jackowski J, Krafft T, Neves M, Divi J, Rasse M, Guerra F, Fischer K. Immediate and early loading of chemically modified implants in posterior jaws: 3-year results from a prospective randomized multicenter study. Clin Implant Dent Relat Res. 2013 Aug;15(4):600-12. doi: 10.1111/j.1708-8208.2011.00418.x. Epub 2011 Dec 15. PMID 22171722

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: From the 280 patients (146/134 immediate/early loading group) who received a study implant 266 patients (138/128 immediate/early loading group) fulfilled all primary and secondary inclusion/exclusion criteria after Implantation. The main effectiveness analysis was performed on this population
Groups:
- Immediate Loading: Implant(s) will be restored with a temporary restoration on the day of surgery
  SLActive dental implant
- Early Loading: Healing caps will be placed on the implant(s) immediately after surgery. A provisional restoration will be placed between day 28 to day 34 post surgery
  SLActive dental implant
Period: Overall Study
Arm/Group | Immediate Loading | Early Loading
Started | 146 | 134
20-23 Weeks | 135 | 124
1 Year | 131 | 120
Surgery (Baseline) (Includes patients who fulfilled all eligibility criteria and received a study implant) | 138 | 128
Completed | 124 | 115
Not Completed | 22 | 19
Not completed — Lost to Follow-up | 2 | 2
Not completed — Withdrawal by Subject | 2 | 1
Not completed — complications | 3 | 1
Not completed — others | 7 | 9
Not completed — not eligible | 8 | 6

BASELINE CHARACTERISTICS:
Population: missing at least one tooth in the posterior maxilla or mandible
Groups:
- Total: Total of all reporting groups
Arm/Group | Immediate Loading | Early Loading | Total
Number analyzed (Participants) | 138 | 128 | 266
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.1 (13.3) | 46.6 (12.4) | 46.3 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 74 | 148
  Male | 64 | 54 | 118
implant distribution maxilla, mandible [Number; unit: participants]
  patients with implants in the maxilla | 47 | 37 | 84
  patients with implants in the mandible | 72 | 79 | 151
  patients with implants in both jaws | 19 | 12 | 31
Number of implants placed [Number; unit: implants] | 197 | 186 | 383

OUTCOME MEASURES:

1. Primary Outcome: Evaluation of Changes in Crestal Bone Levels Evaluated From Standardized Periapical X-rays Comparing the Immediate and Delayed Loading Procedures in Each Group.
Time Frame: Change in crestal bone level from surgery (baseline) to 20-23 Weeks post-surgery
Population: This analysis was based on bone level measurements of implants as observational unit. The final number of units analyzed for the defined period is based on x-rays available at both time points (baseline and follow-up visit). Our statistical analysis of the study data included how many implants were analyzed but not how many participants.
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Implants
Arm/Group | Immediate Loading | Early Loading
Number analyzed (Participants) | NA | NA
Number analyzed (Implants) | 169 | 152
mm | 0.82 (0.89) | 0.56 (0.73)

2. Primary Outcome: Evaluation of Changes in Crestal Bone Levels Evaluated From Standardized Periapical X-rays Comparing the Immediate and Delayed Loading Procedures in Each Group.
Time Frame: Change in crestal bone level from surgery (baseline) to 1 year post-surgery
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Implants
Arm/Group | Immediate Loading | Early Loading
Number analyzed (Participants) | NA | NA
Number analyzed (Implants) | 168 | 155
mm | 0.90 (0.90) | 0.59 (0.79)

3. Primary Outcome: Evaluation of Changes in Crestal Bone Levels Evaluated From Standardized Periapical X-rays Comparing the Immediate and Delayed Loading Procedures in Each Group.
Time Frame: Change in crestal bone level from surgery (baseline) to 2 years post-surgery
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Implants
Arm/Group | Immediate Loading | Early Loading
Number analyzed (Participants) | NA | NA
Number analyzed (Implants) | 157 | 149
mm | 0.89 (0.90) | 0.57 (0.83)

4. Primary Outcome: Evaluation of Changes in Crestal Bone Levels Evaluated From Standardized Periapical X-rays Comparing the Immediate and Delayed Loading Procedures in Each Group.
Time Frame: Change in crestal bone level from surgery (baseline) to 3 years post-surgery
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Implants
Arm/Group | Immediate Loading | Early Loading
Number analyzed (Participants) | NA | NA
Number analyzed (Implants) | 155 | 140
mm | 0.88 (0.82) | 0.57 (0.84)

5. Secondary Outcome: Implant Survival
Description: Implant survival: An implant was deemed to be surviving, if it was still in place at the time of evaluation
Time Frame: 20-23 Weeks post-surgery
Measure: Number; unit: implants
Units Other Than Participants: Implants
Arm/Group | Immediate Loading | Early Loading
Number analyzed (Participants) | 138 | 128
Number analyzed (Implants) | 197 | 186
implants | 193 | 180

6. Secondary Outcome: Implant Survival
Description: Implant survival: An implant was deemed to be surviving, if it was still in place at the time of Evaluation
Time Frame: 1 year post-surgery
Population: Number of implants placed. Implants from drop-outs are not included
Measure: Number; unit: implants
Units Other Than Participants: Number of implants
Arm/Group | Immediate Loading | Early Loading
Number analyzed (Participants) | 138 | 128
Number analyzed (Number of implants) | 197 | 186
implants | 193 | 180

7. Secondary Outcome: Implant Survival
Description: Implant survival: An implant was deemed to be surviving, if it was still in place at the time of Evaluation
Time Frame: 2 years post-surgery
Measure: Number; unit: implants
Units Other Than Participants: Number of Implants
Arm/Group | Immediate Loading | Early Loading
Number analyzed (Participants) | 138 | 128
Number analyzed (Number of Implants) | 197 | 186
implants | 192 | 180

8. Secondary Outcome: Implant Survival
Description: Implant survival: An implant was deemed to be surviving, if it was still in place at the time of Evaluation
Time Frame: 3 years post-surgery
Measure: Number; unit: implants
Units Other Than Participants: Number of Implants
Arm/Group | Immediate Loading | Early Loading
Number analyzed (Participants) | 138 | 128
Number analyzed (Number of Implants) | 197 | 186
implants | 192 | 180

9. Secondary Outcome: Nature and Frequency of Adverse Events (AEs) - Number of Patients Affected
Description: Patients affected by AE Patients affected by related/ unknown AE
Time Frame: until the 3 year post-surgery
Population: All patients who had signed the informed consent form and received a study implant, regardless if all primary and secondary inclusion/exclusion criteria after Implantation were fulfilled
Measure: Number; unit: patients affected
Arm/Group | Immediate Loading | Early Loading
Number analyzed (Participants) | 146 | 134
patients affected
  Patients affected by AE | 38 | 35
  Patients affected by related/ unknown AE | 20 | 15

10. Secondary Outcome: Implant Success
Description: Implant success: An implant was deemed to be successful if there was a lack of implant mobility, absence of any continuous peri-implant radiolucency based on radiographic findings, absence of any recurrent peri-implant infection, absence of continuous or recurrent pain and absence of structural failure of the implant
Time Frame: 20-23 weeks post-surgery
Measure: Number; unit: implants
Units Other Than Participants: Number of Implants
Arm/Group | Immediate Loading | Early Loading
Number analyzed (Participants) | 135 | 124
Number analyzed (Number of Implants) | 191 | 180
implants | 187 | 174

11. Secondary Outcome: Implant Success
Description: as for outcome 10
Time Frame: 1 years post-surgery
Measure: Number; unit: implants
Units Other Than Participants: Number of Implants
Arm/Group | Immediate Loading | Early Loading
Number analyzed (Participants) | 131 | 120
Number analyzed (Number of Implants) | 190 | 178
implants | 185 | 172

12. Secondary Outcome: Implant Success
Description: as for outcome 10
Time Frame: 2 years post-surgery
Population: The analysis was based on implants as observational unit. The 2-year data was analyzed together with the 3-year data. Our statistical analysis for 2-year time point included how many implants were available but not how many participants.
Measure: Number; unit: implants
Units Other Than Participants: Number of Implants
Arm/Group | Immediate Loading | Early Loading
Number analyzed (Participants) | NA | NA
Number analyzed (Number of Implants) | 183 | 172
implants | 177 | 164

13. Secondary Outcome: Implant Success
Description: as for outcome 10
Time Frame: 3 years post-surgery
Measure: Number; unit: implants
Units Other Than Participants: Number of Implants
Arm/Group | Immediate Loading | Early Loading
Number analyzed (Participants) | 124 | 115
Number analyzed (Number of Implants) | 180 | 170
implants | 174 | 164

14. Secondary Outcome: Nature and Frequency of Adverse Events (AEs) - Number of Adverse Events
Description: Number of Adverse Events Number of related/unknown AE Number of related/unknown SAEs Number of Serious Adverse Events (SAEs)
Time Frame: until the 3 year post-surgery
Population: as for outcome 9
Measure: Number; unit: number of events
Arm/Group | Immediate Loading | Early Loading
Number analyzed (Participants) | 146 | 134
number of events
  Number of Adverse Events | 56 | 41
  Number of related/unknown AEs | 26 | 17
  Number of related/unknown SAEs | 0 | 0
  Number of Serious Adverse Events | 3 | 1

ADVERSE EVENTS:
Time Frame: 3 years
Groups:
- Immediate Loading: SLActive Implant(s) will be restored with a temporary restoration on the day of surgery.
- Early Loading: Healing caps will be placed on the SLActive Implant(s) immediately after surgery. A provisional restoration will be placed between day 28 to day 34 post surgery
Arm/Group | Immediate Loading | Early Loading
Serious Adverse Events (participants affected / at risk) | 2/146 | 1/134
Other Adverse Events (participants affected / at risk) | 20/146 | 12/134
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Immediate Loading (N=146) | Early Loading (N=134)
CORNEAL ULCER (Eye disorders) | 1 (2) | 0 (0) — DUE TO PSEUDOMONAS AEGUINOSA INFECTION or PSEUDOMONAS AERGINOSA
stomach canser (Gastrointestinal disorders) | 1 (1) | 0 (0)
PERI - IMPLANT INFECTION (Infections and infestations) | 0 (0) | 1 (1) — not of the study implant
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Immediate Loading (N=146) | Early Loading (N=134)
Prosthetic related complication (Surgical and medical procedures) | 13 (16) | 12 (15) — Failure, fracture, lost of provisional crown. Recementation. Excess of cement removal
Pain, discomfort (General disorders) | 7 (9) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No